CLINICAL TRIAL: NCT06483503
Title: A Prospective Cohort Study Evaluating a Novel Colonoscope With a 230-degree Extra-wide Field of View Optics (EFOV)
Brief Title: Extra Wide Field of View Lens Study
Acronym: EFOV
Status: Active, not recruiting | Type: Observational
Sponsor: Pentax Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CA-PE-EFOV-2024-001 - V1.0
Record Dates: First submitted 2024-06-18; First posted 2024-07-03 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: EFOV Colonoscope — Routine colonoscopy using the EFOV lens in the colonoscope.

SUMMARY:
The goal of this observation study is to learn about the feasibility of a new colonoscope which provides the physician an extra-wide field of view during a screening colonoscopy. The main question this study aims to answer is can this new type of colonoscope locate polyps during clinical use in patients.

Patients will undergo a routine colonoscopy for colorectal cancer or polyp surveillance and have one follow-up phone call up to 2 weeks of the colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Screening for colorectal cancer at the age greater than or equal to 50 years, or evaluation of a positive stool test (i-FOBT) or polyp surveillance.
* Signed informed consent.

Exclusion Criteria:

* ASA classification ≥3.
* Age <18 years.
* Known or suspicion of inflammatory bowel disease.
* Known polyp(s) for polypectomy.
* High risk for colorectal cancer, history of extensive polyposis, patients with known genetic disease.
* Prior colorectal surgery.
* Vulnerable subjects or subjects unable to follow the procedures of the investigation, e.g., due to language problems.
* Unable or unwilling to undergo bowel cleansing for colonoscopy.
* Female patients who are pregnant or nursing.
* Participation in another clinical trial within 30 days prior to the Screening Visit or during this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults scheduled for screening colonoscopies, evaluation of a positive stool test or polyp surveillance colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2024-12-08 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Cecal Intubation Rate | Day 1
  The proportion of procedures in which the cecum was reached.

SECONDARY OUTCOMES:
Procedure Time | Day 1
  Total procedure time and separated into cecal insertion time, time to reach ileum and withdrawal time.
Ileum Intubation Rate | Day 1
  Success rate of reaching the Ileum.
Therapeutic Intervention Success Rate | Day 1
  The ability to collect a biopsy or remove a polyp.
Mean number of polyps per coloscopy and its detection rate | Day 1
  Count of number of polyps seen during colonoscopy
Mean number of adenomas and its detection rate | Day 14
  Count of number of adenomas/sessile serrate lesions defined by pathology
Mean number of sessile serrate lesions and its detection rate | Day 14
  Count of number of adenomas/sessile serrate lesions defined by pathology
Patient Satisfaction Survey | Day 14
  During a follow-up phone call, the patient will be asked a yes or no question to rate their satisfaction of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Horst Neuhaus, MD, PhD, Principal Investigator — RKM 740 Interdisciplinary Specialist Clinic
Locations (1):
- RKM 740 Interdisciplinary Care Clinic - Gastroenterology, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: No